CLINICAL TRIAL: NCT04614675
Title: Transarticular Lateral Release Versus Percutaneous Lateral Release in Combination With Distal Metatarsal Chevron Osteotomy for Hallux Valgus -A Prospective Randomized Controlled Trial-
Brief Title: Transarticular Lateral Release Versus Percutaneous Lateral Release for Hallux Valgus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-07-021B
Record Dates: First submitted 2020-07-19; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Hallux Valgus
Keywords: Hallux valgus; Distal soft tissue procedure; Transarticular lateral release (TALR); Percutaneous lateral release (PCLR); Minimally invasive surgery
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transarticular lateral release (TALR) (Active Comparator): TALR The first toe is pulled distally for access into the lateral aspect of first MTPJ. A No.15 beaver blade is advanced from the medial incision laterally to divide the lateral capsule vertically and adductor hallucis tendon. Same intraoperative stress test is performed and recorded under fluoroscope to confirm correction.
  Interventions: Procedure: Distal soft tissue procedure with TALR
- Percutaneous lateral release (PCLR) (Active Comparator): PCLR A 0.5 cm stab wound is made at lateral aspect of first MTPJ. A No. 15 beaver blade is advanced into the lateral side of MTPJ with a quarter of the blade inside the joint and verified with fluoroscope. The blade is turned laterally to face the adductor hallucis tendon. The adductor tendon is divided with lateral movement of the blade and varus manipulation of proximal phalanx. A click is heard as adequate release of adductor hallucis tendon. Same intraoperative stress test is performed and recorded under fluoroscope to confirm correction.
  Interventions: Procedure: Distal soft tissue procedure with PCLR

INTERVENTIONS:
Procedure: Distal soft tissue procedure with TALR — TALR group: Transarticular lateral release as the distal soft tissue procedure
  Arms: Transarticular lateral release (TALR)
Procedure: Distal soft tissue procedure with PCLR — PCLR: Percutaneous soft tissue procedures as the distal soft tissue procedure
  Arms: Percutaneous lateral release (PCLR)

SUMMARY:
background Hallux valgus (HV) is a common forefoot disorder in need of surgical intervention after failed conservative treatment. Surgical treatment of HV generally includes different kinds of osteotomy in combination with different distal soft tissue procedures (DSTP). Commonly used DSTP are open first-web lateral release, transarticular lateral release (TALR), and percutaneous lateral release (PCLR). In some studies, TALR showed similar surgical outcomes with open first-web space lateral release. Besides, PCLR has been described with satisfactory outcomes. TALR and PCLR are gaining popularity due to their less invasive approach and potential in combination with a distal metatarsal Chevron osteotomy (DMCO). Currently, there is no study comparing the surgical results between TALR and PCLR for surgical reconstruction of HV.

Aim The aim of this prospective randomized trial is to compare the surgical outcomes of TALR versus PCLR, both in combination of DMCO, for the treatment of HV. Our hypothesis is that TALR would achieve a better surgical outcomes than PCLR.

DETAILED DESCRIPTION:
This study will be conducted from January, 2021 to December, 2024. A total of 140 participants are included with 70 participants in each group. Participants are allocated to TALR or PCLR group before index surgery according to a computer-generated randomization list.

For all patients, after regional nerve block and adequate sedation, intraoperative stress test is performed for flexibility of first metatarsophalangeal joint (MTPJ).6 The test is confirmed with dorsoplantar fluoroscopy. Only the cases with negative results (passive correction is not possible) are included. Then, a medial incision of 2.5-cm is made at distal metatarsal head and a reverse L-shaped medial capsulotomy is made followed by TALR or PCLR.

After TALR or PCLR, medial bunionectomy is performed. DMCO is made with the apex at distal metatarsal neck and angle of 60 to 90 degrees. The metatarsal head is laterally moved and fixed with one or 2 oblique headless compression screws.

Postoperative followup The patients are followed up at two weeks for removal of stitches, then 1-month, 2-month, 3-month, 6-months, 1-year, and annually after 1 year for radiographic , functional assessments, and evaluation of complications.

Power analysis for patient number With the assumption of mean HVA are 10 degrees for TALR group and 15 degrees for PCLR group at final followup, and a standard deviation of 8 degrees for both groups, the calculated effect size d is 0.625. In order to achieve the α error probability of 0.05 and power of 0.95, 68 participants in each group are necessary with a total of 136 participants in this study.

Statistical analysis In the comparisons between TALR and PCLR groups, the independent two samples t-test and the Mann-Whitney test are performed for normal and non-normal distributed data respectively, and the Fisher's exact test is performed for categorical data. P-values less than 0.05 is considered to be statistical significant. The statistical analyses are performed by using SPSS 25.0 statistics software (SPSS Inc, Chicago, USA).

Clinical relevance

1. Compare the differences of surgical outcomes between TALR and PCLR. These results could offer valuable information for foot and ankle surgeon.
2. If PCLR is not adequate to achieve satisfactory outcomes, the minimally invasive surgery using PCLR for HV is not recommended.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or greater than 20 years
* Hallux valgus angle (HVA) equal or greater than 20 degrees
* Persistent symptoms after failed conservative treatment
* Receiving DMCO for HV

Exclusion Criteria:

* Underlying rheumatoid or other inflammatory arthritis
* Hallux rigidus
* Recurrent hallux valgus after previous surgery
* First tarsometatarsal hypermobility
* A positive intraoperative stress test for lateral soft tissue release

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
hallux valgus angle (HVA)(degrees) | postoperative 1-month
  weightbearing dorsoplantar radiograph, angle between proximal phalanx and 1st metatarsal
hallux valgus angle (HVA)(degrees) | postoperative 2-month
  weightbearing dorsoplantar radiograph, angle between proximal phalanx and 1st metatarsal
hallux valgus angle (HVA)(degrees) | postoperative 3-month
  weightbearing dorsoplantar radiograph, angle between proximal phalanx and 1st metatarsal
hallux valgus angle (HVA)(degrees) | postoperative 6-month
  weightbearing dorsoplantar radiograph, angle between proximal phalanx and 1st metatarsal
hallux valgus angle (HVA)(degrees) | postoperative 12-month
  weightbearing dorsoplantar radiograph, angle between proximal phalanx and 1st metatarsal
hallux valgus angle (HVA)(degrees) | postoperative 24-month
  weightbearing dorsoplantar radiograph, angle between proximal phalanx and 1st metatarsal
hallux valgus angle (HVA)(degrees) | postoperative 36-month
  weightbearing dorsoplantar radiograph, angle between proximal phalanx and 1st metatarsal
intermetatarsal angle (IMA) 1-2 (degrees) | postoperative 1-month
  weightbearing dorsoplantar radiograph, angle between 1st metatarsal and 2nd metatarsal
intermetatarsal angle (IMA) 1-2 (degrees) | postoperative 2-month
  weightbearing dorsoplantar radiograph, angle between 1st metatarsal and 2nd metatarsal
intermetatarsal angle (IMA) 1-2 (degrees) | postoperative 3-month
  weightbearing dorsoplantar radiograph, angle between 1st metatarsal and 2nd metatarsal
intermetatarsal angle (IMA) 1-2 (degrees) | postoperative 6-month
  weightbearing dorsoplantar radiograph, angle between 1st metatarsal and 2nd metatarsal
intermetatarsal angle (IMA) 1-2 (degrees) | postoperative 12-month
  weightbearing dorsoplantar radiograph, angle between 1st metatarsal and 2nd metatarsal
intermetatarsal angle (IMA) 1-2 (degrees) | postoperative 24-month
  weightbearing dorsoplantar radiograph, angle between 1st metatarsal and 2nd metatarsal
intermetatarsal angle (IMA) 1-2 (degrees) | postoperative 36-month
  weightbearing dorsoplantar radiograph, angle between 1st metatarsal and 2nd metatarsal
sesamoid position | postoperative 1-month
  weightbearing dorsoplantar radiograph, the location of the medial sesamoid with progressive lateral subluxation from grade one to seven according to the classification system of Hardy and Clapham
sesamoid position | postoperative 2-month
  weightbearing dorsoplantar radiograph, the location of the medial sesamoid with progressive lateral subluxation from grade one to seven according to the classification system of Hardy and Clapham
sesamoid position | postoperative 3-month
  weightbearing dorsoplantar radiograph, the location of the medial sesamoid with progressive lateral subluxation from grade one to seven according to the classification system of Hardy and Clapham
sesamoid position | postoperative 6-month
  weightbearing dorsoplantar radiograph, the location of the medial sesamoid with progressive lateral subluxation from grade one to seven according to the classification system of Hardy and Clapham
sesamoid position | postoperative 12-month
  weightbearing dorsoplantar radiograph, the location of the medial sesamoid with progressive lateral subluxation from grade one to seven according to the classification system of Hardy and Clapham
sesamoid position | postoperative 24-month
  weightbearing dorsoplantar radiograph, the location of the medial sesamoid with progressive lateral subluxation from grade one to seven according to the classification system of Hardy and Clapham
sesamoid position | postoperative 36-month
  weightbearing dorsoplantar radiograph, the location of the medial sesamoid with progressive lateral subluxation from grade one to seven according to the classification system of Hardy and Clapham
visual analogue scale (VAS) for pain | postoperative 3-months
  pain score, (0-10, the lower the better)
visual analogue scale (VAS) for pain | postoperative 6-months
  pain score, (0-10, the lower the better)
visual analogue scale (VAS) for pain | postoperative 12-months
  pain score, (0-10, the lower the better)
visual analogue scale (VAS) for pain | postoperative 24-months
  pain score, (0-10, the lower the better)
visual analogue scale (VAS) for pain | postoperative 36-months
  pain score, (0-10, the lower the better)
hallux-metatarsophalangeal-interphalangeal scale of American Orthopaedic Foot Ankle Society (AOFAS) | postoperative 3-months
  functional score, 0-100, the higher the better
hallux-metatarsophalangeal-interphalangeal scale of American Orthopaedic Foot Ankle Society (AOFAS) | postoperative 6-months
  functional score, 0-100, the higher the better
hallux-metatarsophalangeal-interphalangeal scale of American Orthopaedic Foot Ankle Society (AOFAS) | postoperative 12-months
  functional score, 0-100, the higher the better
hallux-metatarsophalangeal-interphalangeal scale of American Orthopaedic Foot Ankle Society (AOFAS) | postoperative 24-months
  functional score, 0-100, the higher the better
hallux-metatarsophalangeal-interphalangeal scale of American Orthopaedic Foot Ankle Society (AOFAS) | postoperative 36-months
  functional score, 0-100, the higher the better

SECONDARY OUTCOMES:
rate of osteonecrosis of first metatarsal head | 12-month
  postoperative complications
rate of osteonecrosis of first metatarsal head | 24-month
  postoperative complications
rate of osteonecrosis of first metatarsal head | 36-month
  postoperative complications
rate of numbness of hallux | 12-month
  postoperative complication
rate of numbness of hallux | 24-month
  postoperative complication
rate of numbness of hallux | 36-month
  postoperative complication
rate of infection | 12-month
  postoperative complication
rate of infection | 24-month
  postoperative complication
rate of infection | 36-month
  postoperative complication
rate of first MTPJ arthritis | 12-month
  postoperative complication
rate of first MTPJ arthritis | 24-month
  postoperative complication
rate of first MTPJ arthritis | 36-month
  postoperative complication
rate of recurrent hallux valgus | 12-month
  postoperative complication, hallux valgus angle equal or greater than 20 degrees
rate of recurrent hallux valgus | 24-month
  postoperative complication, hallux valgus angle equal or greater than 20 degrees
rate of recurrent hallux valgus | 36-month
  postoperative complication, hallux valgus angle equal or greater than 20 degrees
rate of hallux varus | 12-month
  postoperative complication
rate of hallux varus | 24-month
  postoperative complication
rate of hallux varus | 36-month
  postoperative complication
rate of reoperations | 12-month
  postoperative complication
rate of reoperations | 24-month
  postoperative complication
rate of reoperations | 36-month
  postoperative complication

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Ching Chiang, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagner E, Ortiz C, Figueroa F, Vela O, Wagner P, Gould JS. Role of a Limited Transarticular Release in Severe Hallux Valgus Correction. Foot Ankle Int. 2015 Nov;36(11):1322-9. doi: 10.1177/1071100715593082. Epub 2015 Jul 7. PMID 26152873
- [Background] Lee KB, Cho NY, Park HW, Seon JK, Lee SH. A comparison of proximal and distal Chevron osteotomy, both with lateral soft-tissue release, for moderate to severe hallux valgus in patients undergoing simultaneous bilateral correction: a prospective randomised controlled trial. Bone Joint J. 2015 Feb;97-B(2):202-7. doi: 10.1302/0301-620X.97B2.34449. PMID 25628283
- [Background] Park CH, Jang JH, Lee SH, Lee WC. A comparison of proximal and distal chevron osteotomy for the correction of moderate hallux valgus deformity. Bone Joint J. 2013 May;95-B(5):649-56. doi: 10.1302/0301-620X.95B5.30181. PMID 23632675
- [Background] Park YB, Lee KB, Kim SK, Seon JK, Lee JY. Comparison of distal soft-tissue procedures combined with a distal chevron osteotomy for moderate to severe hallux valgus: first web-space versus transarticular approach. J Bone Joint Surg Am. 2013 Nov 6;95(21):e158. doi: 10.2106/JBJS.L.01017. PMID 24196470
- [Background] Ahn JY, Lee HS, Chun H, Kim JS, Seo DK, Choi YR, Kim SW. Comparison of open lateral release and transarticular lateral release in distal chevron metatarsal osteotomy for hallux valgus correction. Int Orthop. 2013 Sep;37(9):1781-7. doi: 10.1007/s00264-013-2023-1. Epub 2013 Aug 6. PMID 23917851
- [Background] de Las Heras-Romero J, Lledo-Alvarez AM, Andres-Grau J, Picazo-Marin F, Moreno-Sanchez JF, Hernandez-Torralba M. A new minimally extended distal Chevron osteotomy (MEDCO) with percutaneous soft tissue release (PSTR) for treatment of moderate hallux valgus. Foot (Edinb). 2019 Sep;40:27-33. doi: 10.1016/j.foot.2019.04.001. Epub 2019 Apr 4. PMID 31055210
- [Background] Lucas y Hernandez J, Golano P, Roshan-Zamir S, Darcel V, Chauveaux D, Laffenetre O. Treatment of moderate hallux valgus by percutaneous, extra-articular reverse-L Chevron (PERC) osteotomy. Bone Joint J. 2016 Mar;98-B(3):365-73. doi: 10.1302/0301-620X.98B3.35666. PMID 26920962
- [Background] Bock P, Kluger R, Kristen KH, Mittlbock M, Schuh R, Trnka HJ. The Scarf Osteotomy with Minimally Invasive Lateral Release for Treatment of Hallux Valgus Deformity: Intermediate and Long-Term Results. J Bone Joint Surg Am. 2015 Aug 5;97(15):1238-45. doi: 10.2106/JBJS.N.00971. PMID 26246258
- [Background] Kim HN, Suh DH, Hwang PS, Yu SO, Park YW. Role of intraoperative varus stress test for lateral soft tissue release during chevron bunion procedure. Foot Ankle Int. 2011 Apr;32(4):362-7. doi: 10.3113/FAI.2011.0362. PMID 21733437
- [Background] Choi YR, Lee HS, Jeong JJ, Kim SW, Jeon IH, Lee DH, Lee WC. Hallux valgus correction using transarticular lateral release with distal chevron osteotomy. Foot Ankle Int. 2012 Oct;33(10):838-43. doi: 10.3113/FAI.2012.0838. PMID 23050706
- [Background] Dalmau-Pastor M, Malagelada F, Cordier G, Del Vecchio JJ, Ghioldi ME, Vega J. Anatomical Study of Minimally Invasive Lateral Release Techniques for Hallux Valgus Treatment. Foot Ankle Int. 2020 Aug;41(8):984-992. doi: 10.1177/1071100720920863. Epub 2020 May 26. PMID 32456480
- [Background] Okuda R, Kinoshita M, Yasuda T, Jotoku T, Kitano N, Shima H. Postoperative incomplete reduction of the sesamoids as a risk factor for recurrence of hallux valgus. J Bone Joint Surg Am. 2009 Jul;91(7):1637-45. doi: 10.2106/JBJS.H.00796. PMID 19571086